CLINICAL TRIAL: NCT04175301
Title: Pilot Study on Effects of Hydrogen Rich Water on Quality of Life of Patients Treated With Radiotherapy for High Grade Gliomas.
Brief Title: Effect H2 Water on QoL of Patients Receiving Radiotherapy for High Grade Gliomas.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Agnieszka Kowalska, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2019-00236
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Malignant Glioma
Keywords: neuroprotection; hydrogen; antioxidant; malignant glioma
MeSH Terms: conditions — Glioma | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects will be randomly assigned in a 2:1 ratio to receive hydrogen or placebo, additionally to all standard-of-care treatments by the SB Research Pharmacy. Masking of active and placebo treatments will be preserved by creating study medication containers that appear identical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrogen (Experimental): Five times per day for 6 weeks subjects will dissolve a hydrogen generating tablet into water and drink the effervescent water. Dissolving one tablet in 250 mL of water will achieve a saturating hydrogen concentration of approximately 1.6 ppm.
  Interventions: Drug: Hydrogen
- Placebo (Placebo Comparator): Five times per day for 6 weeks subjects will dissolve an placebo tablet into water and drink the effervescent water. The effervescent placebo tablet does not generate hydrogen-enriched water.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydrogen — Each hydrogen tablet contains 80 mg magnesium
  Other Names: H2
  Arms: Hydrogen
Drug: Placebo oral tablet — Matching placebo tablet also contains 80 mg magnesium
  Arms: Placebo

SUMMARY:
This is a pilot randomized control trial (RCT) to explore the effects of hydrogen rich water on quality of life in patients with high grade gliomas, receiving focal radiation therapy to the brain concurrent with chemotherapy with Temozolomide.

DETAILED DESCRIPTION:
This will be a pilot trial exploring the ability of molecular hydrogen to improve quality of life in patients with high grade gliomas, receiving focal radiation therapy to the brain concurrent with chemotherapy with Temozolomide. Hydrogen has an excellent safety profile, has antioxidant properties and reduces inflammatory events in the tissues. It has been postulated in previous studies that continuous consumption of hydrogen water reduces oxidative stress in the brain by lowering the concentration of the reactive oxygen species, resulting in the improvement of adult neurogenesis or the stimulation of neural proliferation, leading to the prevention of the decline in the learning and memory.

This will be a double blinded, placebo-controlled trial. Eligible and willing subjects will be randomly assigned in a 2:1 ratio to be treated with either hydrogen or placebo, to receive hydrogen or placebo, additionally to all standard-of-care treatments. The treatment with hydrogen or placebo will start the day before chemoradiation therapy starts, and continue for six weeks. The effects of drinking hydrogen water on the quality of life will be assessed using the EORTC QLQ-C30 and the EORTC QLQ-BN20 questionnaires at baseline, at 6 weeks, 6 months, 12 months, 18 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or over
* New diagnosis of a malignant glioma (HGG) either by a biopsy or craniotomy
* KPS of at least 70
* Being able to fill out quality of life questionnaire

Exclusion Criteria:

* Other major diseases of the central nervous system, including history of prior brain tumors, Alzheimer's disease, Parkinson's disease, demyelinating disease, inflammatory brain or vascular disease, traumatic encephalopathy, or idiopathic intracranial hypertension, anxiety/depression.
* Pre-existing neurological disability, unable to read or write
* Severe comorbidities likely to result in patient dying within 3 months
* Prior history of head/neck radiation therapy
* Other active cancer or history of other cancer diagnosed within 5 year.
* Inability to safely tolerate the 1500 ml- 2000ml fluid load (po water) associated with study medication*
* Pregnancy or nursing.
* Treatment with another investigational drug within the last 30 days that may interfere with this study's medications*
* Hypersensitivity to Temozolomide and or it's active agent- Dacarbazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient enrollment statistics | 3 years
  Feasibility of recruitment, assessment procedures, treatment, and outcome measures will be evaluated. Number of screened / eligible / enrolled patients, treatment adherence, assessment completion, subject dropout, data completeness, and data variability.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) C30 score | 2 years
  Change in health related quality of life from baseline to week 6, month 6, month 12, month 18, and month 24, as assessed by the EORTC QLQ-C30 score. The score range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) BN20 score | 2 years
  Change in health related quality of life from baseline to week 6, month 6, month 12, month 18, and month 24, as assessed by the EORTC QLQ-BN20 score. The score range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Memory | 2 years
  Change in memory from baseline to week 6, month 6, month 12, month 18, and month 24, as assessed by the Mini-Mental State Examination (MMSE).
Karnofsky performance score (KPS) | 2 years
  Change in Karnofsky performance score (KPS) from baseline to week 6, month 6, month 12, month 18, and month 24.
Overall survival and progression free survival (PFS) | 2 years
  Overall survival is defined as the time from randomization until death from any cause. PFS is defined as the time from randomization until tumor progression (defined by McDonald's criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Kowalska, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No